CLINICAL TRIAL: NCT06459609
Title: Effect of Protein Supplementation on Craving in Subjects Hospitalised for Addiction Treatment. Monocentric Pilot Study.
Brief Title: Effect of Protein Supplementation on Craving in Subjects Hospitalised for Addiction Treatment
Acronym: CRAVPROT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-A01230-47
Record Dates: First submitted 2024-05-30; First posted 2024-06-14 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Addiction
Keywords: addiction; craving; protein supplementation
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P - SP (Other): 1 week with protein supplementation (P) then one week without protein supplementation (SP)
  Interventions: Dietary Supplement: protein supplementation
- SP - P (Other): 1 week without protein supplementation (SP) then one week with protein supplementation (P)
  Interventions: Dietary Supplement: protein supplementation

INTERVENTIONS:
Dietary Supplement: protein supplementation — Protein supplementation takes the form of a powder sachet mixed with yoghurt or compote. It will be given twice a day, at the same time.

SUMMARY:
Moncentric pilot study conducted in the addictology department of the Pau Hospital, designed to demonstrate the benefit of protein supplementation on craving in patients with a substance use disorder at the start of their treatment for addiction.

This study will be conducted according a crossover design with a one-week phase with protein supplementation (P) and a one-week phase without protein supplementation (SP).

DETAILED DESCRIPTION:
Addiction is a chronic psychiatric disorder characterised by the loss of control over the use of rewarding substances or behaviours, despite the accumulated damage. Craving, defined as an irrepressible, obsessive craving, is a key early symptom of addiction. Protein supplementation could reduce this craving. Nutritional abnormalities aggravate addictions but no study have directly assessed the impact of protein supplementation on craving. Evidence suggests that protein supplementation reduces cravings for sugary and hyperpalatable foods, which could extend to rewarding substances. The hypothesis is that this supplementation reduces the intensity, duration and frequency of craving in withdrawal patients by influencing dopaminergic reward circuits.

Protein supplementation takes the form of a powder sachet mixed with yoghurt or compote. It will be given twice a day, at the same time (8am and 4pm).

Patients will be enrolled at the admission to the addiction unit. They will be assessed psychologically, addictologically and nutritionally for one week and then will be randomised. Patients will be asked to assess their cravings, dietary needs, consumption of addictive substances and palatable foods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Aged 18 and over
* Admitted for complex care in the addictology department
* Person affiliated to or benefiting from a social security scheme
* Free, informed and written consent signed by the participant and the investigator

Exclusion Criteria:

* Allergy to milk protein
* Admitted to hospital for less than 3 weeks
* Severe somatic or psychiatric pathology incompatible with understanding assessment tools
* Difficulty understanding and/or writing French
* Presumed non-compliant in completing the patient diary
* Person participating in another research study with an exclusion period still in progress
* Person under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of craving for the main substance | This outcome will be assessed twice a day (morning and afternoon) from day 8 to day 21, during the period with and without protein supplementation.
  Evaluation of the evolution of craving for the main substance in patients with a substance use disorder in association with protein supplementation. It will be a self-assessment by the patient, using a visual analogue craving scale ranging from 1 'no craving' to 7 'extreme craving'.

SECONDARY OUTCOMES:
Food craving evolution | This outcome will be assessed twice a day (morning and evening) from Day 8 to Day 21 during the period with and without protein supplementation.
  Food craving will be assessed by patient self-assessment using a visual analogue craving scale ranging from 1 'no craving' to 7 'extreme craving'.
Consumption of hyperpalatable foods | This outcome will be assessed every day from Day 8 to Day 21 during the period with and without protein supplementation.
  Consumption of hyperpalatable foods will be assessed by patient self-evaluation, twice a day from D8 to D21 during the period with and without protein supplementation, using a visual scale assessing the extent to which the patient consumed hyperpalatable foods outside of meals, this scale ranging from 1 'not at all' to 7 'very much'.
Influence of the severity of addiction | Evaluation at the inclusion
  Influence of the severity of addiction measured using the Addiction Severity Index (ASI) questionnaire
Influence of psychiatric comorbidities | Evaluation at the inclusion
  Influence of psychiatric comorbidities (mood disorders and anxiety disorders) assessed using the MINI (Mini International Neuropsychiatric Interview)

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Pau, Pau, France

IPD SHARING:
Plan to Share IPD: No